CLINICAL TRIAL: NCT01951742
Title: Dose Finding Study of Botulinum Neurotoxin Type A In Subjects With Crow's Feet (Lateral Canthal Lines)
Brief Title: Dose Finding Study In Subjects With Crow's Feet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterios Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANT-1401-LCL-204
Record Dates: First submitted 2013-09-22; First posted 2013-09-27 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Lateral Canthal Lines; Crow's Feet
Keywords: wrinkles

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Vehicle (Placebo Comparator): vehicle without ANT-1401
  Interventions: Biological: Vehicle
- Dose 1 (Experimental): lowest dose
  Interventions: Biological: ANT-1401
- Dose 2 (Experimental): second lowest dose
  Interventions: Biological: ANT-1401
- Dose 3 (Experimental): mid-level dose
  Interventions: Biological: ANT-1401
- Dose 4 (Experimental): second highest dose
  Interventions: Biological: ANT-1401
- Dose 5 (Experimental): highest dose
  Interventions: Biological: ANT-1401

INTERVENTIONS:
Biological: ANT-1401 — Active
  Arms: Dose 1; Dose 2; Dose 3; Dose 4; Dose 5
Biological: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to establish the therapeutic range of ANT-1401 in the treatment of Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* 30 - 60 years of age
* mild to moderate Crow's Feet wrinkles at rest
* moderate to severe Crow's Feet wrinkles on contraction
* willingness to refrain from any product affecting skin remodeling
* female subjects must be not pregnant and non-lactating

Exclusion Criteria:

* history of peri-ocular surgery, brow lift or related procedures
* procedures affecting the lateral canthal region in the prior 12 months
* application of topical prescription medication to the treatment area
* female subjects who are pregnant or are nursing a child

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Investigators Global Assessment Scale | Week 4
  Crow's Feet Wrinkle Scale

SECONDARY OUTCOMES:
Subject Self-Assessment score | up to 12 12 weeks
  Subjects self assessment of severity of Crow's Feet

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Miami, Florida
  - Pinellas Park, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Rochester, New York
  - High Point, North Carolina
  - Knoxville, Tennessee
  - Norfolk, Virginia